CLINICAL TRIAL: NCT04659811
Title: A Phase II Study of Stereotactic Radiosurgery in Conjunction With the PD-1 Inhibitor, Pembrolizumab for the Treatment of Recurrent Meningioma
Brief Title: Stereotactic Radiosurgery and Immunotherapy (Pembrolizumab) for the Treatment of Recurrent Meningioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Ann Oberheim Bush, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Nancy Ann Oberheim Bush, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19109; NCI-2020-11359 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Grade I Meningioma, Adult; Grade II Meningioma, Adult; Grade III Meningioma, Adult; Recurrent Meningioma
Keywords: PD-1 Inhibitor; Stereotactic Radiosurgery; Immunotherapy; Pembrolizumab
MeSH Terms: conditions — Meningioma | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment for recurrent meningioma (pembrolizumab, stereotactic radiosurgery) (Experimental): Participants with recurrent grade II or III meningioma will receive stereotactic radiosurgery. in conjunction with pembrolizumab 200mg IV infusion on day 1 (to -1) of radiation and then every 3 weeks. Participants may be eligible for up to 17 additional cycles of pembrolizumab depending on disease status after completion of first course.
  Interventions: Drug: Pembrolizumab; Procedure: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Pembrolizumab — 200mg given intravenously (IV) on day 1 (to -1) of radiation and then every 3 weeks until progression or unacceptable toxicity
  Other Names: Keytruda; Pembrolizumab IV
Procedure: Stereotactic Radiosurgery — Given in (a) single session treatment with margin dose of 15-20 Gy to the target for a maximum target volume of 8 cc or (b) five consecutive business days treatment to total dose of 25-30 Gy to the target for a maximum target volume of 20 cc when the target volume exceeds 8 cc or the target is in proximity to critical structures
  Other Names: SRS

SUMMARY:
This phase II trial studies the effect of stereotactic radiosurgery and pembrolizumab in treating patients with meningioma that has come back (recurrent). Stereotactic radiosurgery is a type of external radiation therapy that uses special equipment to position the patient and precisely give a single large dose of radiation to a tumor. It is used to treat brain tumors and other brain disorders that cannot be treated by regular surgery. Pembrolizumab is a humanized monoclonal antibody. An antibody is a common type of protein made in the body in response to a foreign substance. Antibodies attack foreign substances and protect against infection. Antibodies can also be produced in the laboratory for use in treating patients; an antibody that is made in the lab is also known as a humanized monoclonal antibody. Pembrolizumab is a highly selective humanized monoclonal antibody that is designed to block the action of the receptor PD-1. It has been studied in lab experiments and in other types of cancer. The PD-1 receptor works to keep the immune system from noticing tumor cells. The addition of pembrolizumab to stereotactic radiosurgery may improve the progression free survival of patients with meningioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of stereotactic radiation and pembrolizumab for treatment of recurrent meningioma compared to historical control based on progression free survival at 12 months (PFS12).

SECONDARY OBJECTIVE:

I. To assess overall survival and further assess progression free survival of stereotactic radiation and pembrolizumab for treatment of recurrent meningioma.

EXPLORATORY OBJECTIVES:

I. To assess immune-related tumor effects pembrolizumab treatment in meningioma using magnetic resonance (MR) imaging in conjunction with assessment by Response Assessment in Neuro-Oncology Criteria (RANO) and Immunotherapy (i)RANO criteria.

II. To assess neurocognitive function and quality of life with pembrolizumab and radiation using the Neurologic Assessment in Neuro-Oncology (NANO) Scale, and European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire brain tumour module (QLQ-BN20).

III. To assess safety of the combined treatment modalities in meningioma, through evaluation of grade III adverse events (AEs) and dose-limiting toxicity (DLT).

OUTLINE:

Within -3 to 0 days from the start of stereotactic radiation therapy, patients receive pembrolizumab intravenously (IV) over 30 minutes on days 1 and 22. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo stereotactic radiosurgery on day 1 or days 1-5 of cycle 1 in the absence of disease progression or unacceptable toxicity.

All participants who have completed the first course, or stopped for complete response, may be eligible for up to an additional 17 cycles of pembrolizumab if there is investigator-determined progressive disease by iRANO after initial treatment.

After completion of study treatment, patients are followed up at 30 days, every 12 weeks for 2 years, and then every 6 months thereafter for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed World Health Organization (WHO) grade II or III meningioma that is progressive or with one or more recurrences following surgical resection and radiotherapy
* Patients must be eligible/appropriate for treatment with radiation therapy, specifically, if radiation is given in a single session, the target volume cannot exceed 8 ccs or if given in five (consecutive business days) sessions, the target volume cannot exceed 20 ccs
* Prior therapy:

  * There is no limit on the number of prior surgeries or systemically administered therapeutic agents
  * An interval of >= 28 days and full recovery (no ongoing safety issues) from surgical resection
  * An interval of > 7 days from stereotactic biopsy
  * For prior systemic agents, participants must be at least 4 weeks (or 5 half-lives, whichever is shorter) from other prior cytotoxic chemotherapy (6 weeks from nitrosoureas) or biologic therapies
  * For prior radiotherapy, there are no exclusions on number of courses or prior type of radiotherapy. All modalities including prior fractionated external beam photon/proton radiotherapy, stereotactic radiosurgery, and/or or brachytherapy are permissible with a required interval of 6 months from last prior radiotherapy treatment, unless radiation given outside of the planned field, then within 2 weeks from prior radiotherapy treatment. Patients must have had one prior course of radiation therapy
* Participants must have recovered to grade =< 1 or pretreatment baseline from clinically significant adverse events related to prior therapy (excluding alopecia, laboratory values listed per inclusion criteria and lymphopenia)
* Be >= 18 years of age on day of signing informed consent
* Have a Karnofsky performance status (KPS) >= 70
* Absolute neutrophil count (ANC) >= 1500/microliter (uL) (within 28 days prior to enrollment)
* Platelets >= 100000/uL (within 28 days prior to enrollment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (within 28 days prior to enrollment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 28 days prior to enrollment) (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl))

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 28 days prior to enrollment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT)) =< 2.5 x ULN (within 28 days prior to enrollment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (within 28 days prior to enrollment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 28 days prior to enrollment)
* Additional required screening labs within 28 days: albumin, Alkaline phosphatase, calcium, total bilirubin, blood urea nitrogen (BUN), creatinine, total protein, random glucose, potassium, sodium, chloride,bicarbonate, and magnesium, phosphorus.
* Magnetic resonance imaging (MRI) within 28 days prior to start of study drug. Corticosteroid dose must be less than or equal to 2 mg and at a stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI and the start of treatment, a new baseline MRI is required
* Ability to understand and the willingness to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by MRI, as confirmed by signing a written informed consent document
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason:

  * Male participants:

    ** A male participant must agree to use a contraception during the treatment period and for 120 days after the last dose of study treatment and refrain from donating sperm during this period
  * Female participants:

    * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

      * Not a woman of childbearing potential (WOCBP) OR
      * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment

Exclusion Criteria:

* WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Tumors that are primarily localized to the brainstem or spinal cord, NOTE: patients with known tumors in these areas that are not progressive are not excluded
* Known metastasis outside if the central nervous system (CNS), however, no baseline staging is required
* Evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade =< 1 and either post-operative or stable on at least 2 consecutive MRI scans
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137)
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Prior treatment with systemic immunosuppressive treatments, such as methotrexate, chloroquine, azathioprine, etc. within 3 months of start of study therapy
* No concurrent treatment on another clinical trial for 4 weeks (or 5 half-lives, whichever is shorter) for prior systemic agents, other prior cytotoxic chemotherapy (6 weeks from nitrosoureas) or biologic therapies. Supportive care trials or non- treatment trials, e.g. quality of life, are allowed
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Steroids for cerebral edema are allowed if less than or equal to 2 mg of dexamethasone
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) (testing not required)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen (HBsAg) reactive) or known active hepatitis C virus (defined as hepatitis C virus (HCV) ribonucleic acid (RNA) is detected) infection
* Has a known history of active Bacillus tuberculosis (TB)
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Progression Free Survival at 12 months (PFS12) | Up to 12 months
  Percentage of patients who are progression-free at the landmark of 12 months from start of treatment based on the target lesion(s) that are receiving radiation treatment will be reported. Tumor progression will be assessed using Immunotherapy Radiologic Assessment in Neuro-oncology Criteria (iRANO) and defined as > 25% increase in sum of the products of perpendicular diameters of enhancing lesions (over baseline if no decrease) on stable or increasing doses of corticosteroids and/or a significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids compared to baseline scan or best response following initiation of therapy, not due to co-morbid events.

SECONDARY OUTCOMES:
Median overall survival (OS) | Up to 5 years
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death estimated from the Kaplan-Meier method.
Median progression free survival (PFS) | Up to 5 years
  PFS is defined as the duration of time from start of treatment to time of progression using Immunotherapy Radiologic Assessment in Neuro-oncology Criteria (iRANO) or death estimated from the Kaplan-Meier method, and two-sided 95% confidence intervals (CI) will be computed based on the Greenwood's formula.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Oberheim Bush, MD, PhD, Principal Investigator — University of California, San Francisco; Steve Braunstein, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No